CLINICAL TRIAL: NCT03813602
Title: Effects of Cannabis on Driver Performance and Eye Movements and Characteristics During Simulated Driving: Feasibility Study
Brief Title: Detection of Cannabis Impairment With an Eye Tracker
Acronym: ACS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 076/2018
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Cannabis Intoxication
MeSH Terms: interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cannabis sativa (Experimental): a 750 mg cannabis cigarette with 12.5% THC
  Interventions: Drug: Cannabis Sativa

INTERVENTIONS:
Drug: Cannabis Sativa — 750 mg cannabis cigarette with 12.5% THC
  Other Names: Marijuana

SUMMARY:
Cannabis is one of the widely used psychoactive substances in the world. With increasing legalization, the prevalence of driving under the influence of cannabis will undoubtedly rise. At present, roadside detection of cannabis intoxication is largely dependent on drug recognition experts who rely on changes in eye movements when impaired. In this regard, use of eye trackers can help to detect impairment in drivers. The purpose of the present study is to determine the feasibility of the use of eye trackers in detecting impairment in participants who smoked a cannabis cigarette.

DETAILED DESCRIPTION:
Participants will attend one study session after determination of eligibility. During this session, they will smoke a cannabis cigarette with 12.5% THC prior to driving a simulator. Driving will be assessed prior to smoking cannabis and at 7 time points after smoking cannabis. Eye tracking measures will also be taken while driving after smoking cannabis. Blood will be drawn for determination of levels of the psychoactive substance THC and its metabolites. Saliva tests, urine tests and subjective tests will also be performed at various times points after smoking cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Weekly use of cannabis (1 to 4 days per week) confirmed by urine point-of-care testing;
* 19-26 years of age;
* holds a class G or G2 Ontario driver's licence (or equivalent from another jurisdiction) for at least 12 months;
* Willing to abstain from using alcohol for 48 hours and cannabis for 72 hours prior to the study session;
* Willing to abstain from all other drugs not prescribed for medical purposes for the duration of the study;
* Provides written and informed consent.

Exclusion Criteria:

* Urine toxicology screens negative for cannabis upon eligibility assessment;
* Diagnosis of severe medical or psychiatric conditions;
* Females: Pregnancy or breastfeeding;
* Meets criteria for Alcohol or Substance Dependence (current or lifetime) (DSM-IV);
* Is a regular user of medications that affect brain function (i.e., antidepressants, benzodiazepines, stimulants);
* First-degree relative diagnosed with schizophrenia.

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in eye gaze | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Measures of eye movement with an eye tracker

SECONDARY OUTCOMES:
Change in saccades | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Measures of quick eye movements with an eye tracker
Change in eye fixations | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Measure of where the eye is looking with an eye tracker
Change in blinking rate | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The number of blinks, measured with an eye tracker
Change in blinking duration | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The length of time that blinks last, measured with a eye tracker
Change in blinking speed | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  How fast the blinking is, measured with an eye tracker
Change in pupil size | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The diameter of pupils while driving, measured with an eye tracker
Change in mean speed on the driving simulator | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The speed, in km, while driving a driving simulator
Change in standard deviation of speed on the driving simulator | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The amount of variation in speed while driving the driving simulator
Change in maximum speed on the driving simulator | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The greatest speed obtained on the driving simulator
Change in standard deviation of lateral position on the driving simulator | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The amount of weaving while driving the driving simulator
Change in minimum time to collision on the driving simulator | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The time needed to collide with the car in front, while driving the simulator
Change in number of collisions | baseline, 15 minutes, 35 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The number of times a car impacts another car while driving the simulator
Change in blood concentrations of delta-9-tetrahydrocannabinol | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The levels of the psychoactive component of cannabis, THC, in blood
Change in blood concentrations of carboxy-tetrahydrocannabinol | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The levels of the inactive metabolite of THC in blood
Change in blood concentrations of 11-hydroxy-tetrahydrocannabinol | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The levels of the active metabolite of THC in blood
Change in saliva THC detection | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Detection of THC in saliva
Change in systolic blood pressure | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Vital signs
Change in diastolic blood pressure | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Vital signs
Change in heart rate | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Vital signs
Change in temperature | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Vital signs
Change in number of respirations per minute | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  Vital signs
Change in Subjective cannabis effects with a visual analog scale | baseline, 5 minutes, 25 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours
  The amount of liking of cannabis from 0 to 100, with 100 being the greatest value

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD PhD, Principal Investigator — Centre for Addition and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shahidi Zandi A, Comeau FJE, Mann RE, Di Ciano P, Arslan EP, Murphy T, Le Foll B, Wickens CM. Preliminary Eye-Tracking Data as a Nonintrusive Marker for Blood Delta-9-Tetrahydrocannabinol Concentration and Drugged Driving. Cannabis Cannabinoid Res. 2021 Dec;6(6):537-547. doi: 10.1089/can.2020.0141. Epub 2021 Aug 24. PMID 34432541